CLINICAL TRIAL: NCT00026130
Title: A Phase II Trial of Gemcitabine, 5-Fluorouracil and Radiation Therapy in Locally Advanced Non-Metastatic Pancreatic Adenocarcinoma
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-80003; U10CA031946 (NIH); CALGB-80003; CDR0000068988 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + 5FU + XRT (Experimental): Chemo and radiation therapy in the treatment of non-metastatic pancreatic cancer
  Interventions: Drug: fluorouracil; Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: fluorouracil — 200mg/sq m/d CIVI 5/7 days during radiation therapy (wks 1-6)
  Other Names: 5FU
Drug: gemcitabine hydrochloride — 200mg/sq m IV infusion over 30 min wkly (on d 1, 2, OR 3) during radiation tx (wks 1-6) 1000mg/sq m IV infusion over 30 min wkly for 3 weeks during ea chemotherapy cycle
Radiation: radiation therapy — 4500cGy total in 25 fractions M-F followed by 540cGy in 3 fractions (Total dose 5040cGy)during radiation tx (wks 1-6)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and radiation therapy in treating patients who have locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival of patients with locally advanced non-metastatic pancreatic adenocarcinoma treated with gemcitabine, fluorouracil, and radiotherapy.
* Determine the time to progression in patients treated with this regimen.
* Determine the overall clinical response in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes once weekly and fluorouracil IV continuously on days 1-5 weekly for 6 weeks. Patients concurrently undergo radiotherapy 5 days a week for 6 weeks.

Three weeks after the completion of chemoradiotherapy, patients receive gemcitabine IV over 30 minutes once weekly on weeks 1-3. Treatment repeats every 4 weeks for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 78 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic adenocarcinoma

  * Non-metastatic disease that is unresectable due to any of the following:

    * Tumor greater than 5 cm
    * Bulky lymph nodes greater than 2 cm, but within the radiation port
    * Vascular involvement or impingement of major vessels
    * Involvement of colon, adrenal glands, or kidney
* Measurable or evaluable disease
* No prior therapy for pancreatic adenocarcinoma
* No peritoneal seeding or other evidence of metastatic disease by laparotomy or laparoscopy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* CTC 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months

Other:

* No other uncontrolled serious medical or psychiatric illness that would preclude study compliance
* No other malignancy within the past 5 years except limited or curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* No prior abdominal radiotherapy

Surgery:

* At least 2 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2001-09; Primary Completion 2005-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 9 months up to 3 years post treatment

SECONDARY OUTCOMES:
Time to progression | After 2 cycles of tx, then q 2 mon for 1 yr then q 3 mon for 2 yrs
Clinical Response | q 2 mon for Yr 1 post Tx, then q 3 mon for 2 yrs
CA19-9 Levels | q cycle, then q 2 mon for 1 yr, then q 3 mon for 2 yrs
  Biomarker response
Toxicity | q cycle

CONTACTS AND LOCATIONS:
Overall Officials: Harvey J. Mamon, MD, PhD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center
Locations (77):
- United States (77):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Mamon HJ, Niedzwiecki D, Hollis DR, et al.: Preliminary analysis of Cancer and Leukemia Group B (CALGB) 80003: a phase II trial of gemcitabine, 5-fluorouracil (5FU), and radiation therapy (RT) in locally advanced non-metastatic pancreatic adenocarcinoma. [Abstract] Int J Radiat Oncol Biol Phys 63 (Suppl 1): A-22, S13, 2005.